CLINICAL TRIAL: NCT04784663
Title: Public Messaging to Increase Treatment Seeking Among Veterans at Risk for Suicide During Transition From Military Service
Brief Title: Public Messaging to Increase Treatment Seeking for Veterans at Risk for Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SDR 19-354; HX003130-01A2 (Other Grant/Funding Number: VA Health Services Research & Development)
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Mental Health; Suicide
Keywords: communication; Veterans; public health; treatment engagement
MeSH Terms: conditions — Psychological Well-Being; Suicide; Communication

STUDY DESIGN:
Intervention Model Description: All participants will complete the consent process and baseline assessment by telephone with an RA and are randomized to receive the intervention at either baseline (T1), 1-month (T2) or 2-month follow up (T3). Exposure to intervention occurs over a 1-month period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Message Exposure (Experimental): Participants exposed to 4 study videos over a one-month period and complete telephone-based assessments at baseline, 1- and 2-month follow up. Study videos are delivered by study's mobile app downloaded to participants' own Smartphone.
  Interventions: Behavioral: Messaging
- Wait List Control (Placebo Comparator): While wait-listed, participants will receive one push notification each week thanking them for participation, informing them that they will receive messages in the near future or reminding them of the length of the study. Telephone-based assessments are completed at baseline, 1- and 2-month follow up. Push notifications are delivered by study's mobile app downloaded to participants' own Smartphone.
  Interventions: Other: Wait list control

INTERVENTIONS:
Behavioral: Messaging — Four brief video messages, each approximately 1.5 minutes in length, focused on facilitating treatment seeking by addressing barriers and improving attitudes. Intervention delivered to participant by study mobile app downloaded to participants' own smartphone.
  Arms: Message Exposure
Other: Wait list control — one push notification each week thanking individuals for participation, informing them that they will receive messages in the near future or reminding them of the length of the study.
  Arms: Wait List Control

SUMMARY:
The risk for suicide increases by nearly 50% in the first year that service members transition from the military to civilian life underscoring the need for effective strategies to facilitate help seeking among Veterans vulnerable to self-directed violence. Yet despite a great need for treatment, more than half of returning Veterans at risk for suicide do not initiate mental health services. VA has embarked on the regular use of communication campaigns as part of a public health approach designed to reach the larger Veteran population with messages promoting help seeking. However, what types of messages effectively change beliefs and behaviors for at-risk Veterans resistant to seek treatment is unclear. The main objective of this study is to develop and test the use of public messaging to increase treatment seeking among Veterans at risk for suicide and resistant to seek mental health care following separation from military service. This represents the first study to systematically develop public messaging strategies for populations at risk for suicide.

DETAILED DESCRIPTION:
The main objective of this study is to develop and test the use of public messaging to increase treatment seeking among Veterans at risk for suicide and resistant to seek mental health care following separation from military service. A four-year mixed methods study that uses a sequential embedded design will be used to collect data from nationwide samples of Veterans at risk for suicide not in mental health treatment who separated from the DoD in the past year. Informed by the Theory of Planned Behavior, individual interviews will first be conducted to guide the design of effective public messages that will be subsequently tested in a two-arm RCT to determine exposure effects among targeted audience vs. control group. Messages will be disseminated to study participants during the trial by a smartphone app. Research staff will collect assessments by telephone at baseline, 1- and 3-months post-randomization. Potential participants (for all study aims) will be identified using data available from the VA/DOD Identity Repository (VADIR) and recruited by invitational mailing and follow-up telephone calls. If the intervention is found effective, the investigators will work with the VA operational partner to include messages in future outreach approaches to prevent Veteran suicide and use findings to improve current communication performance measures.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran that separated from military service in the past 12 months (any discharge type);
* >18 years old;
* experiencing suicidal ideation;
* low intent to seek help;
* capable of understanding the goals of the study;
* willing and able to provide verbal consent; and 7) smartphone ownership and willing to download/use study mobile app

Exclusion Criteria:

* currently (or in the past 12 months) in formal mental health treatment services;
* deemed impaired during eligibility screening; and 3) currently institutionalized

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
change in treatment initiation from baseline to 1- and 2-month follow-up | baseline, 1-month and 2-month follow up
  change in treatment initiation (yes/no)

SECONDARY OUTCOMES:
change in beliefs about mental health and treatment seeking from baseline to 1- and 2-month follow-up | baseline, 1-month and 2-month follow up
  Change in level of agreement with the following beliefs (a) attitudes toward treatment, (b) subjective norm, (c) perceived behavioral control over treatment is measured using a 7-point likert scale (7 indicating strong agreement)
change in intentions to seek treatment from baseline to 1- and 2-month follow-up | baseline, 1-month and 2-month follow up
  change in intent to seek mental health treatment in the next month measured using a 7-point likert scale (7 indicating strong intent)
change in perceived treatment barriers from baseline to 1- and 2-month follow-up | baseline, 1-month and 2-month follow up
  change in level of agreement with barriers to mental health care that impede one's own behaviors measured using a response scale from 1 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Karras-Pilato, PhD, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (1):
- VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only a Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.

DOCUMENTS (1):
  • Informed Consent Form (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04784663/ICF_000.pdf